CLINICAL TRIAL: NCT03012542
Title: Randomized Trial of Diet for Crohn's Disease and Impact on Disease Activity and the Microbiome
Brief Title: Diet as Essential Therapy (DIET) for Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Timothy Zisman, Associate Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00003247
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet 1 (Experimental): Administered for 8 weeks.
  Interventions: Dietary Supplement: Diet 1
- Diet 2 (Experimental): Administered for 8 weeks.
  Interventions: Dietary Supplement: Diet 2

INTERVENTIONS:
Dietary Supplement: Diet 1 — Diet controlled in amount and source of carbohydrates or fiber containing foods.
  Arms: Diet 1
Dietary Supplement: Diet 2 — Diet controlled in amount and source of carbohydrates or fiber containing foods.
  Arms: Diet 2

SUMMARY:
Recent data suggest that diet in inflammatory bowel disease (IBD) may lead to both symptom control and disease remission. Historically certain diets have been recommended for patients with Crohn's disease during exacerbations despite lack of data supporting efficacy. The investigators propose to evaluate two such diets by randomizing 32 subjects with mildly to moderately active Crohn's disease to one of two diets that differ in the amount and type of carbohydrates and fiber. Subjects will remain on the diet for 8 weeks and will be evaluated for changes from baseline in inflammatory biomarkers, symptomatic disease activity, and the microbiome.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to receive one of two diets that are thought to be beneficial for Crohn's disease for a period of 8 weeks.

Initial evaluation will include a clinic visit with physical exam, medication review, supplemental documentation, and labs. Patients will be asked about their food allergies and intolerances against a master list of all ingredients used in both diets. Patients will then be provided with instructions on how to record their baseline dietary intake for two weeks prior to the intervention diet.

At day 0 patients will begin their study diet. All study meals will be provided to the subject and an approved snack list for the randomized diet will be provided in a sealed envelope with their first week of meals.

At the conclusion of intervention patients will be asked to resume their previous diet for 4 weeks and record their dietary intake. Stool and blood will be collected at baseline and at 4, 8, and 12 weeks. At the conclusion of the study patients will be told which diet they were on and will be provided with dietary consultation by a registered dietitian.

Subjects who withdraw from the study before the 4 week assessment will be asked to provide a final stool sample at the time of withdrawal. If more than 2 subjects drop out prior to week 4, subject replacement will occur.

ELIGIBILITY:
Inclusion Criteria:

* Consentable adults of age 18 or older.
* Diagnosis of Crohn's disease made by a primary gastroenterologist based upon history, physical exam, laboratory/radiological studies, and endoscopy with biopsy.
* Fecal Calprotectin ≥ 300
* Mild to moderate disease activity based upon a modified Harvey Bradshaw Index score of 5-16.
* On stable medication doses for ≥ 2 months.

Exclusion Criteria:

* Inability/unwillingness to adhere to dietary recommendations.
* Allergy or intolerance to any major component of the diets. Major component defined as an ingredient which, when left out of intervention diets, may affect study outcomes.
* Allium intolerance
* Exclusively vegetarian diet
* Active intra-abdominal or perianal abscess/fistula
* Symptomatic bowel stricture
* Other serious medical conditions such as neurological, liver, kidney, autoimmune, or systemic disease
* Use of corticosteroids within 1 month prior to baseline visit
* Tobacco, alcohol, or illicit drug abuse
* Pregnant subjects
* Celiac disease
* Patients already on one of the diets being studied
* C. difficile or other enteric infection (O&P, stool enterics)
* Antibiotic use within 2 months prior to baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Fecal Calprotectin Remission | 8 weeks
  To compare the proportion of patients with calprotectin remission (fecal calprotectin level < 250 and a decrease by ≥ 100 points) at 8 weeks post-dietary intervention for subjects on each diet

SECONDARY OUTCOMES:
Fecal Calprotectin Response | 8 weeks
  Calprotectin response (decrease by ≥ 100 points) or calprotectin improvement (decrease by > 50%) at weeks 4 and 8 for subjects on each diet. Comparison of the mean calprotectin between the 2 treatment groups.
Clinical Response | 8 weeks
  Proportion of patients on each diet with clinical response (HBI score decrease by ≥ 3) or remission (HBI score < 5) at weeks 4 and 8
Metagenomics | 8 weeks
  To compare changes in the metagenomics of the fecal microbiome at 8 weeks relative to baseline for each diet
Microbiota correlation with clinical disease activity and inflammatory biomarkers | 8 weeks
  To determine if changes in the microbiota are associated with changes in clinical disease activity (HBI score), or inflammatory biomarkers (fecal calprotectin, C-reactive protein, etc.).
Future Use | 8 weeks
  To collect stool and blood for potential future analysis looking at proteomics and metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Zisman, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests from investigators will be evaluated on a case by case basis. Data that may be shared include lab values, patient reported outcomes, questionnaires, and microbiome sequences. Specimens may also be shared. Researchers can request data from the study's Principal Investigator in writing.

REFERENCES:
- [Background] Hou JK, Abraham B, El-Serag H. Dietary intake and risk of developing inflammatory bowel disease: a systematic review of the literature. Am J Gastroenterol. 2011 Apr;106(4):563-73. doi: 10.1038/ajg.2011.44. PMID 21468064
- [Background] Richman E, Rhodes JM. Review article: evidence-based dietary advice for patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2013 Nov;38(10):1156-71. doi: 10.1111/apt.12500. Epub 2013 Sep 17. PMID 24102340
- [Background] Wu GD, Chen J, Hoffmann C, Bittinger K, Chen YY, Keilbaugh SA, Bewtra M, Knights D, Walters WA, Knight R, Sinha R, Gilroy E, Gupta K, Baldassano R, Nessel L, Li H, Bushman FD, Lewis JD. Linking long-term dietary patterns with gut microbial enterotypes. Science. 2011 Oct 7;334(6052):105-8. doi: 10.1126/science.1208344. Epub 2011 Sep 1. PMID 21885731
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Manichanh C, Borruel N, Casellas F, Guarner F. The gut microbiota in IBD. Nat Rev Gastroenterol Hepatol. 2012 Oct;9(10):599-608. doi: 10.1038/nrgastro.2012.152. Epub 2012 Aug 21. PMID 22907164